CLINICAL TRIAL: NCT05846581
Title: Observational Prospective Post-Market Clinical Follow-Up (PMCF) Registry of GORE® ACUSEAL Vascular Graft in Dialysis Access
Brief Title: Registry of GORE® ACUSEAL Vascular Graft in Dialysis Access
Acronym: AVG22-09
Status: Recruiting | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: AVG 22-09
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Diseases; End Stage Renal Disease on Dialysis
Keywords: Post-Market Clinical Follow-Up; Chronic Kidney Diseases; End Stage Renal Disease; Hemodialysis; vascular graft
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- ESRD patients that require hemodialysis access through the GORE® ACUSEAL Vascular Graft.: Patient population - patients with CKD in ESRD that require hemodialysis access through the GORE® ACUSEAL Vascular Graft.
  Registry subject population - those patients with CKD in ESRD that require hemodialysis access through the GORE® ACUSEAL Vascular Graft meeting the inclusion and exclusion criteria will be eligible for screening for participation in this registry.
  The registry has been designed with broad eligibility criteria to capture real-world GORE® ACUSEAL Vascular Graft use, for which the device is intended to be implanted. Only patients who meet all of the inclusion criteria and none of the exclusion criteria will be implanted.
  No vulnerable populations are included in this registry.
  Interventions: Device: GORE® ACUSEAL Vascular Graft

INTERVENTIONS:
Device: GORE® ACUSEAL Vascular Graft — The device placement will be performed according to each participating site's standard practice. No specific procedures are required by the protocol.
  At the time of the GORE® ACUSEAL Vascular Grafts implantation, procedural and adverse event information will be collected.

SUMMARY:
The goal of this observational study is to evaluate safety and performance of GORE® ACUSEAL Vascular Graft for the treatment of CKD in patients with ESRD in hemodialysis. The main questions it aims to answer are:

* Safety: Freedom from device-related infection adverse events at 24 months from device implant
* Performance: Secondary patency at 24 months from device implant.

Participants, after informed consent is obtained, will be implanted with GORE® ACUSEAL Vascular Graft and followed for 24 months in standard of care, to evaluate safety and performance of the device.

DETAILED DESCRIPTION:
This is a European, Observational, Non-Interventional, Prospective, Non-Randomized, Single Arm, Multicenter, PMCF Registry to evaluate safety and performance of GORE® ACUSEAL Vascular Graft for the treatment of CKD in patients with ESRD in hemodialysis. There is no comparator device.

The aim of study is to obtain real-world observational evidence about the use of the device.

The AVG 22-09 registry consists of End-Stage Renal Disease (ESRD) patients who require hemodialysis access through Vascular Graft per the evaluating physician.

A total of 72 subjects will be implanted in this registry with a limit of 25 subjects implanted per site.

The registry has been designed with standard eligibility criteria to enroll subjects for which the registry device is intended to treat. Only patients who meet all of the inclusion criteria and none of the exclusion criteria will be implanted. All patients must provide informed consent prior to any registry related procedures being performed and the patient is considered enrolled when informed consent is obtained.

The primary objective is to evaluate safety and performance of GORE® ACUSEAL Vascular Graft in hemodialysis access for the treatment of Chronic Kidney Disease (CKD) in patients with End Stage Renal Disease (ESRD).

All patients who sign an informed consent will be considered enrolled and at the completion of study participation, subjects will be advised by their respective clinical centers on the appropriate follow up regimen to be followed but it is expected that the each implanted subject will be evaluated through hospital discharge and return for follow-up visits per site standard of care.

Each enrolled and implanted subject will be followed for 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. The patient requires the creation of vascular access for hemodialysis secondary to a diagnosis of End-Stage Renal Disease and intends to use GORE® ACUSEAL Vascular Graft device for arteriovenous (AV) access.
2. Age ≥18 years at time of Informed Consent Form (ICF) signature.
3. Willingness of the patient to adhere to institutional standard of care follow-up.
4. Informed Consent Form (ICF) is signed by the patient.
5. The patient is currently on hemodialysis or intended to begin hemodialysis immediately following placement of the GORE® ACUSEAL Vascular Graft device or up to 30 days following placement of the device.
6. The patient has a reasonable expectation of remaining on hemodialysis for 12 months.

Exclusion Criteria:

1. The patient currently has a known or suspected systemic infection.
2. The patient is pregnant or breastfeeding.
3. The patient had a separate interventional or surgical vascular procedure within the study limb within 30 days prior to treatment with the GORE® ACUSEAL Vascular Graft device.
4. The patient had a previous documented (via imaging technique) and unsuccessfully treated ipsilateral central venous stenosis.
5. The patient is currently taking maintenance corticosteroids and immunosuppressant medication such as rapamycin, mycophenolate or mycophenolic acid, prednisone (> 10 mg), cyclosporine, tacrolimus, or cyclophosphamide.
6. The patient has a known hypercoagulability or bleeding disorder.
7. The patient has had a previous instance of Heparin Induced Thrombocytopenia type 2 (HIT-2) or has known sensitivity to Heparin.
8. The patient is enrolled in an investigational study.
9. The patient has been previously enrolled in this registry.
10. The patient is currently being considered for a live donor kidney transplant (living donor either related or unrelated to patient).
11. The patient has life expectancy less than 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Registry subject population - those patients with CKD in ESRD that require hemodialysis access through the GORE® ACUSEAL Vascular Graft meeting the inclusion and exclusion criteria will be eligible for screening for participation in this registry.
  The registry has been designed with broad eligibility criteria to capture real-world GORE® ACUSEAL Vascular Graft use, for which the device is intended to be implanted. Only patients who meet all of the inclusion criteria and none of the exclusion criteria will be implanted.
  No vulnerable populations are included in this registry.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2027-10-27 (Estimated); Study Completion 2027-10-27 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint. Number of subjects free from device-related infection at 24 months from device implant. | 24 months from device implant
  Events will be computed as follows:
  1. All subjects who had a registry device related AE with an Infection MedDRA code within 730 days from device implant will be tabulated as 'Not Free from Infection'.
  2. All subjects who completed the registry and were infection free at 24 months from the registry procedure will be considered free from device related infection.
  All relevant infection MedDRA terms will be agreed upon by the Office of Medical Affairs within Gore. This endpoint will be treated as a patient-based binomial proportion, and no formal hypothesis will be tested. A Kaplan Meir analysis will also be done to account for censoring.
Primary Performance Endpoint. Secondary Patency at 24 months: The time from device implant to complete abandonment of the access site for hemodialysis regardless of the number of interventions required to restore or maintain patency. | 24 months from device implant
  Events will be computed as follows:
  1. All subjects who have an abandonment or explant of the registry graft within 730 days will have lost secondary patency. The date will be noted on the discontinuation form.
  2. All subjects who completed the registry within 730 days without a graft abandonment will be considered patent.
  3. If a subject did not complete the registry for a reason other than graft abandonment or explant, they will be censored.
  A Kaplan Meir analysis will be done to account for censoring.

SECONDARY OUTCOMES:
Percentage of GORE® ACUSEAL Vascular Grafts cannulated within 1, 2, 3, 7, and 14 days from device implant. | Cannulation within 1, 2, 3, 7 and 14 days from device implant.
  The percentage of GORE® ACUSEAL Grafts cannulated within 24, 48,72,168, and 336 hours post device implant will be computed as follows:
  1. The hours from end time of procedure to the first successful hemodialysis session performed through the GORE® ACUSEAL Graft will be recorded per subject.
  This endpoint will be treated as a patient-based binomial proportion and will be summarized as percent with a 95% confidence interval.
Percentage of Subjects free from bleeding events through 6, 12, and 24 months from device implant. | 6, 12, and 24 months from device implant
  1. All subjects experiencing an adverse event classified as bleeding prior to the end of the designated window will be counted as having a bleeding event within that interval.
  2. Subjects not experiencing case 1, who have had a follow-up visit after the beginning of the designated interval, are declared as having no bleeding event.
  3. All subjects not experiencing case 1 or 2 will not be included in computations for the corresponding interval. A Kaplan Meir analysis will be done to account for censoring.
Secondary Patency at 6 and 12 months: The time from device implant to complete abandonment of the access site for hemodialysis regardless of the number of interventions required to restore or maintain patency. | 6 and 12 months from device implant.
  Events will be computed as follows:
  1. All subjects who have an abandonment or explant of the registry graft within 730 days will have lost secondary patency. The date will be noted on the discontinuation form.
  2. All subjects who completed the registry within 730 days without a graft abandonment will be considered patent.
  3. If a subject did not complete the registry for a reason other than graft abandonment or explant, they will be censored.
  A Kaplan Meir analysis will be done to account for censoring.
Primary patency at 6, 12 and 24 months from device implant. Time interval of uninterrupted patency from device implant to the next access thrombosis or intervention. | 6, 12 and 24 months from device implant.
  Primary Patency will be calculated at 6 months, 12 months, and 24 months from device implant, and will use the following decision rules:
  1. Subjects who have a repeat intervention, thrombosis event, abandonment or explant of the registry graft prior to the end of the analysis window will have lost patency.
  2. Subjects who have not experienced case 1, and had a follow-up visit within the desired analysis window are considered patent.
  3. All other subjects will be censored.
  A Kaplan Meir analysis will be done to account for censoring.

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Tozzi, Principal Investigator — University of Insubria (Italy)
Locations (5):
- Germany (2):
  - Evangelisches Klinikum Bethel (EvKB), Bielefeld
  - Ev. DiakonissenKrankenhaus Leipzigemeinnützige, Leipzig
- ASST-Settelaghi Ospedale di Circolo e Fondazione Macchi, Varese, Italy
- United Kingdom (2):
  - North Bristol NHS Trust Southmead Hospital, Bristol, England
  - King's College Hospital NHS Foundation Trust, London, England